CLINICAL TRIAL: NCT06198478
Title: Tandem: Skin-to-skin Transfer From the Delivery Room to the Neonatal Unit for Neonates Above 1500 g
Brief Title: Tandem: Skin-to-skin Transfer From the Delivery Room to the Neonatal Unit
Acronym: Tandem
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2019/510
Record Dates: First submitted 2023-11-30; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-11

CONDITIONS: Preterm Birth; Neonatal Respiratory Distress; Mother-Infant Interaction
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immediate skin-to-skin contact (SSC) is already standard care for healthy term newborns, but its use for term or preterm newborns requiring admission to neonatal unit (NICU) with or without respiratory support is challenging. This study aimed to assess the safety and feasibility of SSC during the transfer of newborn infants, using a new purpose-built mobile shuttle care-station, called "Tandem".

A monocentric prospective observational study was conducted at the tertiary referral center of the Université libre de Bruxelles in Brussels, Belgium Infants born with a birth weight above 1500g were eligible. Following initial stabilization, infants were placed in SSC with one of their parents and transferred to the NICU using the Tandem.

DETAILED DESCRIPTION:
Prior to delivery, the trained neonatal team prepares both the Tandem and a transport incubator as a backup. Delayed umbilical cord clamping will be performed for at least one minute unless prompt resuscitation required. Then, infants will be stabilized on a resuscitation table following European Resuscitation Council guidelines, with applying electrodes for continous monitoring of heart rate, saturation and temperature. After initial stabilization respiratory support will be continued if needed using the Tandem's gas supply. In cases when, antibiotics or continuous IV glucose infusion are necessary, peripheral venous catheters will be placed before departure. In case of respiratory support, nasogastric tube will be insterted. Infants will be then transferred to the NICU under the supervision of a pediatric nurse and/or pediatrician with the Tandem in skin-to-skin position with either the mother or the father. Whenever possible, SSC will be continued for at least 120 minutes before placing the infant in an incubator. Blood glucose measurement will take place at least once during the procedure.

ELIGIBILITY:
Inclusion Criterias:

* neonates with an estimated foetal weight above1500 grams
* neonates requiring admission to the neonatal intensive care unit
* neonates requiring or not non-invasive respiratory support
* neonates with at least one parent who has a good understanding of the method of transfer

Exclusion Criteria:

* neonates presenting a malformation incompatible with this type of transfer
* neonates with invasive ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates over 31 weeks of gestational age and over 1500 grams requiring admission to the neonatal unit
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Skin-to-skin transfer | 0-2 hours of life
  Rate of discontinuation of the skin-to-skin was measured

SECONDARY OUTCOMES:
Safety of Skin-to-skin transfer - Hemodynamic | 0-2 hours of life
  Heart rate measured in bpm (considered normal range: 120-180 bpm )
Safety of Skin-to-skin transfer - Oxygenisation | 0-2 hours of life
  Saturation measured in % ( considered normal >92 %)
Safety of Skin-to-skin transfer- Temperature | 0-2 hours of life
  Temperature measured in Celsius ( considered normal range: 36.5-37.5 C)
Safety of Skin-to-skin transfer - Blood glucose | 0-2 hours of life
  Blood glucose level measured in mg/dL at least once during the first two hours of life (considered normal range: 30-100 mg/dL)
Parental and nursing satisfaction | 0-1 days of life
  Parental and nursing satisfaction with skin-to-skin transfer via the Tandem from the delivery suite or the operating theater to the NICU were rated on a scale from 1 to 10 (10 being the most satisfied)
Breastfeeding at hospital discharge | 1 day (at discharge)
  Exclusive breastfeeding rate at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dorottya KELEN, Principal Investigator — Erasme University Hospital
Locations (1):
- Neonatal Unit Hopital Erasme, Brussels, Anderlecht, Belgium

REFERENCES:
- [Background] Agudelo S, Diaz D, Maldonado MJ, Acuna E, Mainero D, Perez O, Perez L, Molina C. Effect of skin-to-skin contact at birth on early neonatal hospitalization. Early Hum Dev. 2020 May;144:105020. doi: 10.1016/j.earlhumdev.2020.105020. Epub 2020 Mar 25. PMID 32220769
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] van den Berg J, Jakobsson U, Selander B, Lundqvist P. Exploring physiological stability of infants in Kangaroo Mother Care position versus placed in transport incubator during neonatal ground ambulance transport in Sweden. Scand J Caring Sci. 2022 Dec;36(4):997-1005. doi: 10.1111/scs.13000. Epub 2021 May 18. PMID 34008205
- [Background] Sontheimer D, Fischer CB, Buch KE. Kangaroo transport instead of incubator transport. Pediatrics. 2004 Apr;113(4):920-3. doi: 10.1542/peds.113.4.920. PMID 15060247
- [Background] Mitchell AJ, Yates C, Williams K, Hall RW. Effects of daily kangaroo care on cardiorespiratory parameters in preterm infants. J Neonatal Perinatal Med. 2013;6(3):243-9. doi: 10.3233/NPM-1370513. PMID 24246597
- [Background] Nimbalkar SM, Patel VK, Patel DV, Nimbalkar AS, Sethi A, Phatak A. Effect of early skin-to-skin contact following normal delivery on incidence of hypothermia in neonates more than 1800 g: randomized control trial. J Perinatol. 2014 May;34(5):364-8. doi: 10.1038/jp.2014.15. Epub 2014 Feb 20. PMID 24556982
- [Background] Hennequin Y, Grevesse L, Gylbert D, Albertyn V, Hermans S, Van Overmeire B. Skin-to-skin back transfers provide a feasible, safe and low-stress alternative to conventional neonatal transport. Acta Paediatr. 2018 Jan;107(1):163-164. doi: 10.1111/apa.14071. Epub 2017 Oct 2. No abstract available. PMID 28898475
- [Background] Kristoffersen L, Stoen R, Hansen LF, Wilhelmsen J, Bergseng H. Skin-to-Skin Care After Birth for Moderately Preterm Infants. J Obstet Gynecol Neonatal Nurs. 2016 May-Jun;45(3):339-45. doi: 10.1016/j.jogn.2016.02.007. Epub 2016 Apr 7. PMID 27063400
- [Background] Lode-Kolz K, Hermansson C, Linner A, Klemming S, Hetland HB, Bergman N, Lillieskold S, Pike HM, Westrup B, Jonas W, Rettedal S. Immediate skin-to-skin contact after birth ensures stable thermoregulation in very preterm infants in high-resource settings. Acta Paediatr. 2023 May;112(5):934-941. doi: 10.1111/apa.16590. Epub 2022 Nov 18. PMID 36333892
- [Derived] M'Rini M, De Doncker L, Huet E, Rochez C, Kelen D. Skin-to-skin transfer from the delivery room to the neonatal unit for neonates of 1,500g or above: a feasibility and safety study. Front Pediatr. 2024 Mar 20;12:1379763. doi: 10.3389/fped.2024.1379763. eCollection 2024. PMID 38571704